CLINICAL TRIAL: NCT07070687
Title: Transcutaneous Electrical Nerve Stimulation in Nerve-Sparing Radical Hysterectomy: Effects on Bladder Management and Quality of Life in Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weiye Yin, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2207256-18
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer; Postoperative Bladder Dysfunction; Urinary Retention; Pelvic Floor Muscle Weakness; Lower Urinary Tract Symptoms; Recovery of Bladder Function; Improvement in Pelvic Floor Muscle Strength; Enhancement of Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Urinary Retention; Lower Urinary Tract Symptoms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Bladder Management (No Intervention): Control group receiving conventional postoperative bladder care without TENS
- TENS with Standard Management (Experimental): Experimental group receiving standard care plus TENS therapy
  -Real-time electrode adjustment based on feedback Administered using MMK520i device (Degas Intelliance)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Low-frequency electrical stimulation (800Hz) applied at CV2/S3 regions twice daily for 7 days using MMK520i device
  Arms: TENS with Standard Management

SUMMARY:
To evaluate the effects of transcutaneous electrical nerve stimulation (TENS) on bladder management, pelvic floor muscle strength, and quality of life (QoL) in patients undergoing nerve-sparing radical hysterectomy (NSRH) for cervical cancer. A total of 78 NSRH patients during May 2023-May 2024 were divided into conventional catheter management (control group, n = 39) and conventional management + TENS (intervention group, n = 39). Outcomes including urinary retention incidence, postvoid residual urine volume (PVR), catheter indwelling duration, intervention compliance, pelvic floor muscle strength grading, voiding function parameters [first desire to void (FD), bladder compliance (BC), maximum cystometric capacity (MCC)], QoL scores (EORTC QLQ-C30: functional, symptom, and global health domains), and safety were assessed. The intervention group demonstrated significantly lower urinary retention incidence, reduced PVR, and shorter catheter duration versus controls (all P < 0.05). Both groups maintained > 90% intervention compliance (P > 0.05). Post-intervention voiding parameters (FD, BC, MCC) improved more significantly in the intervention group (all P < 0.05), with superior pelvic floor muscle strength grading (P < 0.001). QoL assessment revealed lower functional domain scores and higher symptom/global health scores in the intervention group (all P < 0.001). Safety analysis showed only mild dermal reactions in the intervention group, without significant between-group difference in complication rates (P > 0.05). TENS significantly improves bladder function, pelvic floor muscle strength, and QoL in post-NSRH patients with a favorable safety profile, demonstrating substantial clinical value.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed cervical cancer (FIGO stage IB1-IIA2).
* Scheduled for or completed nerve-sparing radical hysterectomy (NSRH) with pelvic lymphadenectomy.
* Successful indwelling urinary catheter placement within 24 hours postoperatively.
* Age 18-70 years.
* Willing to comply with TENS intervention and follow-up assessments.

Exclusion Criteria:

* Pre-existing neurogenic bladder or urinary tract infection (UTI).
* Severe cardiopulmonary, hepatic, or renal dysfunction.
* Hematologic disorders or systemic infections.
* Contraindications to electrical stimulation (e.g., pacemaker, skin lesions at electrode sites).
* Inability to provide informed consent or complete study procedures.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary retention after catheter removal | Within 7 days post-catheter removal (typically postoperative days 14-21).
  Proportion of patients with postvoid residual urine volume (PVR) >100 mL following initial catheter removal, assessed via bladder ultrasound.

SECONDARY OUTCOMES:
Postvoid residual urine volume (PVR) | Measured immediately after catheter removal and at 1-month follow-up.
  Quantification of residual urine volume (mL) via bladder ultrasound after voiding.
Catheter indwelling duration | Up to 30 days postoperatively.
  Total days from surgery to permanent catheter removal.
Pelvic floor muscle strength grading | At 1-month post-intervention.
  Assessed via vaginal examination using a 6-point scale (Grades 0-V).
Voiding function parameters (FD, BC, MCC) | Pre-intervention and 1-month post-intervention.
  * First desire to void (FD): Volume (mL) at initial urge.
  * Bladder compliance (BC): Δvolume/Δpressure (mL/cmH₂O).
  * Maximum cystometric capacity (MCC): Volume (mL) at strong urge.
Quality of Life (EORTC QLQ-C30 scores) | Pre-intervention and 1-month post-intervention.
  Standardized scores for functional, symptom, and global health domains.

OTHER OUTCOMES:
Safety and adverse events | Throughout the intervention period (7 days) and 1-month follow-up.
  Incidence of complications (UTI, urolithiasis, pain) and TENS-related reactions (erythema, paresthesia).
Intervention compliance | During the 7-day intervention period.
  Proportion of participants completing the full TENS protocol (≥90% sessions).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China